CLINICAL TRIAL: NCT07058324
Title: The Effects of Chicory Root-derived Prebiotic on Mood and Stress Responsiveness in Healthy Adults With Mild to Moderate Levels of Stress and Anxiety: a Randomized, Placebo-controlled, Double-blind, Monocentric, Two-armed Parallel, Prospective Study - The PRIME Study
Brief Title: The Effects of Chicory Root-derived Prebiotic on Mood and Stress Responsiveness in Healthy Adults With Mild to Moderate Levels of Stress and Anxiety
Acronym: PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo-Institute (Industry)
Collaborators: Daacro (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Be01-2025
Record Dates: First submitted 2025-06-02; First posted 2025-07-10 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Stress; Healthy Subjects; Anxiety, Mild to Moderate
Keywords: anxiety; prebiotics
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To reduce potential bias, the study will blind all key parties involved: participants, investigators, and those evaluating the outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic fiber (Experimental): The prebiotic fiber group will receive prebiotic fiber during the 4-week intervention period.
  Interventions: Dietary Supplement: Prebiotic fiber
- Placebo control (Placebo Comparator): The placebo group will receive maltodextrin during the 4-week intervention period.
  Interventions: Dietary Supplement: Placebo control

INTERVENTIONS:
Dietary Supplement: Prebiotic fiber — Chicory root-derived prebiotic fiber
  Arms: Prebiotic fiber
Dietary Supplement: Placebo control — Maltodextrin
  Arms: Placebo control

SUMMARY:
Emerging evidence from preclinical research suggests that prebiotic fibres may play a beneficial role in supporting mental health through modulation of the gut-brain axis-a complex communication network linking the gastrointestinal tract and the central nervous system. Chicory root-derived prebiotic fibre, already well-established for its positive effects on glycaemic control and bowel regularity, has recently shown promise in this context. The present study aims to investigate the mental health benefits of chicory root fibre in a larger and more diverse population, thereby contributing to the growing body of evidence supporting nutritional strategies for mental well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer is healthy at the time of screening.
2. TICS Screening Scale of Chronic Stress (SSCS) score ≥ 6.
3. GAD total score ≥ 5 and ≤ 14 indicating mild to moderate anxiety.
4. Male or female aged ≥18 and ≤ 70 years at the time of screening.
5. Body-Mass-Index (BMI) ≥ 18.5 and ≤ 29.9 kg/m2.
6. Volunteer is able and willing to comply with the study instructions.
7. Volunteer is suitable for participation in the study according to the investigator/study personnel.
8. Voluntary, written informed consent to participate in the study.

Exclusion Criteria:

1. No command of local language.
2. Previously or currently diagnosed neurological or psychiatric disorders.
3. Previous history of renal, hepatic, cardiovascular disease or clinically significant diabetes.
4. Gastrointestinal disorders including irritable bowel syndrome (IBS), inflammatory bowel disease (IBD) or other conditions that might affect the gut environment.
5. Contraindication or allergy to any substance in the verum or placebo product incl. lactose or fructose intolerance.
6. Use of drugs (e.g., antibiotics, aspirin, proton pump inhibitors) influencing gastrointestinal function in the previous 8 weeks before the beginning of intervention.
7. Use of laxatives and labelled pre-and probiotics in the previous 4 weeks before the beginning of intervention.
8. Participation in another study with any investigational product within 30 days of screening or during the study.
9. History of drug (recreational) or alcohol abuse.
10. Use of anti-depressants medication including selective serotonin receptor inhibitors or amitriptyline for 3 months prior to screening.
11. Bowel preparation for investigative procedures in the 4 weeks prior to screening.
12. Surgical resection of any part of the bowel.
13. Pregnant or lactating.
14. Regular smoking.
15. Previous Trier Social Stress Test (TSST) participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Anxiety (STAI-X1, state) | Baseline and after 4 weeks (before and during stress protocol TSST).
  Anxiety as a temporary emotional state will be assessed with State-Trait-Anxiety Inventory (STAI-X1, state). Total scores range from 20-80, with higher scores indicate greater levels of current anxiety.
Anxiety (VAS) | Baseline and after 4 weeks (before and during stress protocol TSST).
  Anxiety as a temporary emotional state will be assessed with 100-mm visual analogue scale (VAS). Higher scores shown in VAS indicating higher levels of anxiety.

SECONDARY OUTCOMES:
Beck's Anxiety Inventory (BAI) | Four weeks.
  Beck's Anxiety Inventory (BAI) will be assessed using a 21-item self-reported questionnaire. Total scores range from 0 to 63, with lower scores indicating lower levels of anxiety.
Beck's Depression Inventory (BDI) | Four weeks.
  Beck's Depression Inventory (BDI) will be assessed using a 21-question self-reported rating inventory in a multiple choice format. Total scores range from 0 to 63, with lower scores indicating lower levels of depression.
Depression Anxiety Stress Scale (DASS) | Four weeks.
  Depression Anxiety Stress Scale (DASS) will be assessed using a 21-item questionnaire that include three scales (depression, anxiety and stress) of which each scale includes 7 items, and responses are rated on a 4-point scale (0-3). Higher scores on each subscale indicate greater symptom severity.
Positive and Negative Affect Schedule (PANAS) | Four weeks.
  Positive and Negative Affect Schedule (PANAS) will be assessed using 20 self-reported measures of 10 positive and negative affect items, respectively. Total scores range from 10 to 50, with higher scores indicating higher levels of positive and negative affects.
Salivary cortisol | Baseline and after 4 weeks (before and during stress protocol TSST).
  Chronic stress, but also anxiety and depression can permanently increase cortisol levels and impair various physical and mental functions.
Blood pressure | Baseline and after 4 weeks (before and during stress protocol TSST).
  Blood pressure (BP, systolic and diastolic) will be measured using an automated blood pressure measurement device (OMRON Medizintechnik).
Gut microbiota | Four weeks.
  Stool samples will be collected for gut microbiota profile analysis.
Dietary intake | Four weeks.
  Dietary intake will be recorded during the study using online dietary assessment tool (MyFood24).
Pulse/heart rate | Baseline and after 4 weeks (before and during stress protocol TSST).
  Pulse/heart rate will be measured through Somno HD eco (Somnomedics), using an ECG and continuous BP measurement based on pulse transit time (PTT)

OTHER OUTCOMES:
Adverse events (AEs) | Through study completion, up to 4 weeks.
  All AEs will be collected in the eCRF. The intensity/severity rating is defined as: 1 = mild (awareness of sign or symptom, but easily tolerated); 2 = moderate (discomfort sufficient to cause interference with normal activities); 3 = severe (incapacitating, with inability to perform normal activities)

CONTACTS AND LOCATIONS:
Overall Officials: Juliane Hellhammer, Ph.D., Principal Investigator — Daacro GmbH & Co. KG
Locations (1):
- daacro GmbH & Co. KG, Trier, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No